CLINICAL TRIAL: NCT03291834
Title: A Study on Sports Participation in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Sports Participation in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JessaH_PedEndo002
Record Dates: First submitted 2017-09-01; First posted 2017-09-25 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
Keywords: type 1 diabetes mellitus; sports; child; adolescent
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
On the basis of a questionnaire the participation at sports activities of children and adolescents with type 1 diabetes mellitus will be studied. The occurrence of hypoglycemia and hyperglycemia will be evaluated, as well as the measures to prevent these complications.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with type 1 diabetes mellitus followed at the pediatric diabetes clinic of the Jessa Hospital

Exclusion Criteria:

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with type 1 diabetes mellitus followed at the pediatric diabetes clinic of the Jessa Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Participation at sports | August 2017
  Detailed description of participation at daily sports in school and outside school
Occurence of hypoglycemia or hyperglycemia | August 2017

SECONDARY OUTCOMES:
Measures taken to prevent hypoglycemia or hyperglycemia | August 2017
  The ingestion of extra carbohydrates to prevent hypoglycemia and/or the administration of extra insulin to prevent hyperglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Guy G Massa, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No